CLINICAL TRIAL: NCT03278106
Title: Phase II Trial of Trifluridine/Tipiracil (FTD/TPI (TAS-102)) in Biliary Tract Cancers
Brief Title: TAS-102 in Treating Advanced Biliary Tract Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1642; NCI-2017-01603 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1642 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Results first posted 2019-10-01 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cholangiocarcinoma; Stage III Gallbladder Cancer AJCC v7; Stage IIIA Gallbladder Cancer AJCC v7; Stage IIIB Gallbladder Cancer AJCC v7; Stage IV Gallbladder Cancer AJCC v7; Stage IVA Gallbladder Cancer AJCC v7; Stage IVB Gallbladder Cancer AJCC v7
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TAS-102) (Experimental): Patients receive trifluridine/tipiracil hydrochloride combination agent TAS-102 orally PO BID on days 1-5 and 8-12. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102 — Given PO
  Other Names: Lonsurf; TAS-102; Trifluridine/Tipiracil

SUMMARY:
This phase II trial studies how well trifluridine/tipiracil hydrochloride combination agent TAS-102 (TAS-102) works in treating participants with biliary tract cancers that have spread to other places in the body. Drugs used in the chemotherapy, such as trifluridine/tipiracil hydrochloride combination agent TAS-102, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of trifluridine/tipiracil hydrochloride combination agent TAS-102 (FTD/TPI [TAS-102]) in patients with refractory cholangiocarcinoma using progression-free survival at 16 weeks.

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of FTD/TPI (TAS-102) in patients with refractory cholangiocarcinoma through adverse event monitoring.

II. Further explore the efficacy of FTD/TPI (TAS-102) in patients with refractory cholangiocarcinoma by overall response rates, progression-free survival, and overall survival.

TERTIARY OBJECTIVES:

I. Determine if circulating tumor cells (CTCs) or cell-free deoxyribonucleic acid (DNA) (cfDNA) at baseline correlates with prognosis or response to therapy.

II. Determine if change in CTCs or cfDNA correlates with efficacy endpoints. III. Determine if different mutational status of the tumor will affect efficacy endpoints.

OUTLINE:

Patients receive trifluridine/tipiracil hydrochloride combination agent TAS-102 orally (PO) twice daily (BID) on days 1-5 and 8-12. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of advanced biliary tract cancers including cancers originating in gallbladder who have received at least one line of systemic anticancer therapy;

  * Note: Patients who have either progressed or intolerant to the prior therapy can be included in this study
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate transaminase (AST) or alanine transaminase (ALT) =< 3 x ULN
* Creatinine =< 1.5 x ULN
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood samples for correlative research purposes

Exclusion Criteria:

* Any of the following:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception for at least 3 months after the last dose of the study drug
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm =< 21 days prior to registration
* Receiving any anticancer therapy for biliary tract cancer =< 21 days prior to registration
* Other active malignancy requiring treatment in =< 6 months prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Mahipal, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (TAS-102)
Started | 28
Completed | 27
Not Completed | 1
Not completed — No protocol treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (TAS-102)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 12
    1 | 15

OUTCOME MEASURES:

1. Primary Outcome: 16-Week Progression-free Survival (PFS) Rate
Description: 16-Week Progression-free survival (PFS) rate is defined as the percentage of patients who are progression-free (stable disease, partial response, or complete response as defined by RECIST v1.1 criteria) at 16 weeks post registration.
Time Frame: 16 weeks
Population: Primary analysis population
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (TAS-102)
Number analyzed (Participants) | 25
percentage of patients | 32.0 [14.9 to 53.5]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR defined as the percentage of patients who experience either a partial response or complete response by the given time point. Complete Response (CR):All of the following must be true: a. Disappearance of all target lesions. b. Each target lymph node must have reduction in short axis to <1.0 cm. Partial Response (PR): At least a 30% decrease in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the BSD.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (TAS-102)
Number analyzed (Participants) | 27
percentage of patients | 0 [0 to 12.8]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS will be estimated using the Kaplan-Meier method. Progression-Free Survival (PFS) is defined as the time from study entry to the first of either disease progression or death from any cause, where disease progression will be determined based on RECIST 1.1 criteria. Patients will be censored at the last disease assessment date. The median PFS and 95% confidence interval will be reported.
Time Frame: Time from study entry to the first of either disease progression or death from any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (TAS-102)
Number analyzed (Participants) | 27
months | 3.8 [2.0 to 5.8]

4. Secondary Outcome: Overall Survival (OS)
Description: OS will be estimated using the Kaplan-Meier method. OS is defined as the time from study entry to death from any cause. Patients will be censored at the date patient was last known to be alive. The median OS and 95% confidence interval will be reported.
Time Frame: Time from study entry to death from any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (TAS-102)
Number analyzed (Participants) | 27
months | 6.1 [4.4 to 11.4]

5. Secondary Outcome: Overall Toxicity Rates (Percentages) for Grade 3 or Higher Adverse Events Considered at Least Possibly Related to Treatment, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (v4)
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Up to 3 years
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (TAS-102)
Number analyzed (Participants) | 27
percentage of patients
  Grade 3 | 48.1
  Grade 4 | 11.1

6. Other Pre Specified Outcome: Change in Circulating Tumor Cells (CTCs) or Cell-free Deoxyribonucleic Acid (DNA) (cfDNA)
Description: Will correlate with efficacy endpoints.
Time Frame: Baseline up to 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Circulating Tumor Cells (CTCs) or Cell-free Deoxyribonucleic Acid (DNA) (cfDNA) Analysis at Baseline
Description: Will determine if CTCs or cfDNA at baseline will correlate with prognosis or response to therapy.
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Mutation Status of the Tumor
Description: Will determine if different mutations status of the tumor will affect efficacy endpoints.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: All patient adverse events are summarized below.
Arm/Group | Treatment (TAS-102)
All-Cause Mortality (participants affected / at risk) | 21/27
Serious Adverse Events (participants affected / at risk) | 10/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (TAS-102) (N=27)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 (2)
Biliary tract infection (Infections and infestations) | 1 (4)
Hepatic infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Blood bilirubin increased (Investigations) | 4 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (TAS-102) (N=27)
Anemia (Blood and lymphatic system disorders) | 25 (83)
Watering eyes (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 22 (66)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (9)
Diarrhea (Gastrointestinal disorders) | 12 (36)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 17 (52)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 9 (11)
Edema limbs (General disorders) | 3 (4)
Fatigue (General disorders) | 27 (93)
Fever (General disorders) | 1 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 5 (7)
Neck edema (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4)
Alkaline phosphatase increased (Investigations) | 6 (9)
Aspartate aminotransferase increased (Investigations) | 4 (6)
Blood bilirubin increased (Investigations) | 4 (5)
Lymphocyte count decreased (Investigations) | 3 (4)
Neutrophil count decreased (Investigations) | 15 (38)
Platelet count decreased (Investigations) | 16 (38)
White blood cell decreased (Investigations) | 12 (20)
Anorexia (Metabolism and nutrition disorders) | 20 (54)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Headache (Nervous system disorders) | 1 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (6)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT03278106/Prot_SAP_000.pdf